CLINICAL TRIAL: NCT05857423
Title: The Comparison of Gentle Human Touch's Effect by Mother and Nurse on Pain Level During Heel Blood Sampling in Preterm Infants
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Istanbul University - Cerrahpasa (Other)
Responsible Party: Principal Investigator, Cansu Avlac, Principal Investigator, Istanbul University - Cerrahpasa
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: IstanbulUCCansuAvlaç0000000001
Record Dates: First submitted 2023-03-25; First posted 2023-05-12 (Actual); Last update posted 2023-05-12 (Actual); Status verified 2023-05

CONDITIONS: Infant, Premature
MeSH Terms: conditions — Premature Birth

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Group (Other): Preterm infants who are applied gentle human touch by nurses
  Interventions: Other: Gentle Human Touch
- Experimental Group (Experimental): Preterm infants who are applied gentle human touch by mother
  Interventions: Other: Gentle Human Touch

INTERVENTIONS:
Other: Gentle Human Touch — Gentle Human Touch procedure has 3 step as follows:
  1. Mother/nurse must wash their hands with antimicrobial soap for 3 minutes before starting Gentle Human Touch procedure.
  2. Next, mother/nurse must warm their hands.
  3. Mother/nurse must place their one hand on the infant's head and the other hand on the lower abdomen that covers the waist and hips of the preterm infant, for 15 minute.

SUMMARY:
This study is an experimental randomized controlled study conducted to compare the effect of gentle human touch applied by mother and nurse on pain level during heel blood sampling in preterm infant. The population of the study consists of preterm infants who stay neonatal intensive care unit of state hospital and whose heels blood sampling will be collected. The number of samples for this study was determined as 40 preterm infants with theoretical power of 95%. This study will be started when the researcher informs the families of preterm infants about the research and receives written and oral consent. The preterm infants were divided into 2 groups of 20 preterm infants, including control group who are applied gentle human touch by nurses and the experimental group who are applied gentle human touch by mothers. In the study, the randomization of the sample group was performed through the website named www.randomizer.org. The researcher records physiological measurements (heart rate and oxygen saturation) and the NIPS score before heel lancing. The gentle human touch procedure will be applied to infants in both groups for 10 minutes and then blood will be drawn from the infants' heels. Intervention assessment (KTA, oxygen saturation, and NIPS) will be done after the preterm infant's heel is pricked. The time will be kept when the needle is pricked and the procedure time will be recorded when the blood collection is finished. The time will be kept as soon as the baby starts to cry and the crying time will be recorded when the crying ends. Evaluation of the NIPS/Neonatal Pain Scale will be done by the researcher and a nurse outside the study. Then, inta-rater reliability will be evaluated. After the blood collection, Gentle Human Touch application will be continued for 5 more minutes. At the end of this period, the heart rate, oxygen saturation and NIPS score will be evaluated again.

DETAILED DESCRIPTION:
The hypotheses of the research are as follows:

* Ho: There is no significant difference between the effect of gentle human touch applied by the mother during heel prick procedure of preterm infants on neonatal pain level (NIPS: Neonatal Infant Pain Scale), heart rate, O2 saturation, and crying time, and the effect of gentle human touch applied by the nurse on pain level.
* H1: The NIPS score of neonates who received gentle human touch from their mother during heel prick procedure of preterm infants will be lower than the neonates who received gentle human touch from the nurse.
* H2: The heart rate of neonates who received gentle human touch from their mother during heel prick procedure of preterm infants will be lower than the neonates who received gentle human touch from the nurse.
* H3: The O2 saturation of neonates who received gentle human touch from their mother during heel prick procedure of preterm infants will be higher than the neonates who received gentle human touch from the nurse.
* H4: The crying time of neonates who received gentle human touch from their mother during heel prick procedure of preterm infants will be shorter than the neonates who received gentle human touch from the nurse.

ELIGIBILITY:
Inclusion Criteria:

* Gestational age between 32 and 36 weeks,
* Birth weight 1200 gr or more,
* APGAR score more than 6 at 5 minute,
* No intracranial hemorrhage higher than Grade II,
* Must have a hemodynamic stability (infants receiving ventilator respiratory support, sepsis, cyanosis and heart disease are not included in the sampling),
* Not taking opiates and sedatives within 4 hour before heel lancing,
* No painful procedure was performed 1 hour ago before heel lancing,

Exclusion Criteria:

* Having a congenital anomalies,
* Having a skin disease,
* Receiving respiratory support with a mechanical ventilator,
* Having a surgical operation,

Ages: 32 Weeks to 36 Weeks | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 40 (Estimated)
Dates: Start 2023-05-10 (Estimated); Primary Completion 2023-12-30 (Estimated); Study Completion 2023-12-30 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in pain on the Neonatal Infant Pain Scale (NIPS) at 5 minutes after the heel lancing | Baseline and 5 minutes after the heel lancing
  This scale, behavioral responses to pain as facial expression, crying, breathing pattern, arms, legs, and alertness are evaluated. The preterm infant get a score between 0-7 and is considered to have pain if it gets a score greater than 3.
  Change=(5 minutes after score- baseline score)